CLINICAL TRIAL: NCT02494622
Title: Alternatives to The Surgical Approach for Giant Spinal Schwannomas: A Clinic Trial
Brief Title: Alternative Treatment of Giant Spinal Schwannomas
Status: Completed | Type: Observational
Sponsor: Gulsah Karaoren (Other Government)
Responsible Party: Sponsor-Investigator, Gulsah Karaoren, MD, Umraniye Education and Research Hospital
Organization: Umraniye Education and Research Hospital (Other Government)
Other Study IDs: GK8
Record Dates: First submitted 2015-06-25; First posted 2015-07-10 (Estimated); Last update posted 2015-07-10 (Estimated); Status verified 2015-07

CONDITIONS: Spinal Cord Neoplasms
MeSH Terms: conditions — Spinal Cord Neoplasms

STUDY DESIGN:
Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Schwannomas are benign tumors that can reach giant sizes. The diagnosis and treatment of these cases differ from those of small schwannomas. The aim of this study was to review the diagnoses and surgical approach characteristics of the giant spinal schwannomas (GSS) of patients who underwent surgery.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with benign spinal schwannoma Sridhar Type III, IV and V

Exclusion Criteria:

* Malign spinal schwannoma
* Sridhar Type I and II

Ages: 16 Years to 76 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients, who underwent surgery for benign spinal schwannoma Sridhar Type III, IV and V (all tumors were larger than 2.5 cm).
Sampling Method: Non-Probability Sample
Enrollment: 18 (Actual)
Dates: Start 2008-01; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Effects of the alternative surgical techniques to the amount of the tumor mass which measured by Nurick Scale | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Said Naderi, Proffesor, Study Chair — Umraniye Education and Research Hospital
Locations (1):
- Gulsah Karaoren, Istanbul, Turkey (Türkiye)

REFERENCES:
- [Background] Samii M, Alimohamadi M, Gerganov V. Surgical Treatment of Jugular Foramen Schwannoma: Surgical Treatment Based on a New Classification. Neurosurgery. 2015 Sep;77(3):424-32; discussion 432. doi: 10.1227/NEU.0000000000000831. PMID 26075309
- [Background] Ohnishi Y, Iwatsuki K, Ohkawa T, Ninomiya K, Moriwaki T, Yoshimine T. Differences between Cervical Schwannomas of the Anterior and Posterior Nerve Roots in Relation to the Incidence of Postoperative Radicular Dysfunction. Asian Spine J. 2015 Apr;9(2):263-70. doi: 10.4184/asj.2015.9.2.263. Epub 2015 Apr 15. PMID 25901239